CLINICAL TRIAL: NCT01227655
Title: Efficacy and Safety of BIA 9-1067 in Idiopathic Parkinson's Disease Patients With "Wearing-off" Phenomenon Treated With Levodopa Plus a Dopa Decarboxylase Inhibitor (DDCI): a Double-blind, Randomised, Placebo-controlled, Parallel-group, Multicentre Clinical Study.
Brief Title: Efficacy and Safety of BIA 9-1067 in Idiopathic Parkinson's Disease Patients.
Acronym: BIPARKII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-91067-302; 2010-022366-27 (EudraCT Number); BIA-91067-302 (Other: Bial - Portela & Cª., S.A.)
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Parkinson's Disease
Keywords: Parkinson; PD; Wearing-off; Levodopa/DDCI
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone; Levodopa; Carbidopa; Benserazide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BIA 9-1067 25 mg once daily (QD). (Experimental): BIA 9-1067, OPC, Opicapone 25 mg once daily (QD).
  Interventions: Drug: BIA 9-1067; Drug: Levodopa; Drug: Carbidopa; Drug: Benserazide
- BIA 9-1067 50 mg once daily (QD). (Experimental): BIA 9-1067, OPC, Opicapone 50 mg once daily (QD).
  Interventions: Drug: BIA 9-1067; Drug: Levodopa; Drug: Carbidopa; Drug: Benserazide
- Placebo (Placebo Comparator): PLC, Placebo
  Interventions: Drug: Placebo; Drug: Levodopa; Drug: Carbidopa; Drug: Benserazide

INTERVENTIONS:
Drug: BIA 9-1067 — Capsules will be used.
  Other Names: Opicapone
  Arms: BIA 9-1067 25 mg once daily (QD).; BIA 9-1067 50 mg once daily (QD).
Drug: Placebo — comparator
  Other Names: placebo; PLC
  Arms: Placebo
Drug: Levodopa
  Other Names: L-Dopa
Drug: Carbidopa — DOPA decarboxylase inhibitor (DDCI)
Drug: Benserazide — DOPA decarboxylase inhibitor

SUMMARY:
Parkinson's disease (PD) is a neurodegenerative disorder of unknown aetiology with an estimated incidence of 4.5-16/100,000 persons/year.

BIA 9-1067 is currently being developed by BIAL (Portela & Cª,S.A.) to be used in addition to L-DOPA (Levodopa) /carbidopa or L-DOPA (Levodopa) / preparations in PD patients. Promising results have been obtained for BIA 9-1067 in previous studies.

DETAILED DESCRIPTION:
This study aims to demonstrate the efficacy and safety of BIA 9-1067 used in addition to L-DOPA/DDCI to control the "wearing-off" phenomenon in patients with PD.

DDCI (DOPA decarboxylase inhibitors): benserazide and carbidopa

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form.
2. Male and female subjects between 30 and 83 years old, inclusive.
3. Diagnosed with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria for at least 3 years.
4. Disease severity Stages I-III (modified Hoehn &Yahr staging) at ON.
5. Treated with L-DOPA/DDCI for at least 1 year with clear clinical improvement.
6. Treated with 3 to 8 daily doses of L-DOPA/DDCI, which can include a slow-release formulation.
7. On a stable regimen of L-DOPA/DDCI and other anti-PD drugs for at least 4 weeks before screening.
8. Signs of "wearing-off" phenomenon (end-of-dose deterioration) for a minimum of 4 weeks before screening with average total daily OFF time while awake of at least 1.5 hours, excluding the early morning pre-first dose OFF, despite optimal anti-PD therapy (based on the investigator's judgment.

Exclusion Criteria:

1. Non-idiopathic PD (atypical parkinsonism, secondary [acquired or symptomatic] parkinsonism, Parkinson-plus syndrome).
2. Dyskinesia disability score >3 in the Unified Parkinson's Disease Rating Scale UPDRS) Sub-section IV A, item 33.
3. Severe and/or unpredictable OFF periods.
4. Treatment with prohibited medication: entacapone, tolcapone, neuroleptics, venlafaxine, MAO inhibitors (except selegiline up to 10 mg/day in oral formulation or 1.25 mg/day in buccal absorption formulation or rasagiline up to 1mg/day), or antiemetics with antidopaminergic action (except domperidone) within the month before screening.
5. Treatment with apomorphine within the month before screening or likely to be needed at any time during the study.
6. Dosage change of concomitant anti-PD medication within 4 weeks of screening.
7. Previous or planned (during the entire study duration, including the OL period)deep brain stimulation.
8. Previous stereotactic surgery (e.g. pallidotomy, thalamotomy) for PD or with planned stereotactic surgery during the study period.
9. Any investigational medicinal product within the 3 months (or within 5 half-lives, whichever is longer) before screening.
10. Any medical condition that might place the subject at increased risk or interfere with assessments.

Ages: 30 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bial - Portela & Cª, S.A., S. Mamede Do Coronado, Portugal

REFERENCES:
- [Derived] Lees AJ, Ferreira J, Rascol O, Poewe W, Rocha JF, McCrory M, Soares-da-Silva P; BIPARK-2 Study Investigators. Opicapone as Adjunct to Levodopa Therapy in Patients With Parkinson Disease and Motor Fluctuations: A Randomized Clinical Trial. JAMA Neurol. 2017 Feb 1;74(2):197-206. doi: 10.1001/jamaneurol.2016.4703. PMID 28027332

RESULTS

PARTICIPANT FLOW:
Groups:
- BIA 9-1067 25 mg; BIA 9-1067 50 mg: BIA 9-1067 once daily (QD).
Period: Overall Study
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | Placebo
Started | 129 | 154 | 144
Safety Set | 125 | 150 | 136
Full Analysis Set | 125 | 147 | 135
Completed | 118 | 128 | 130
Not Completed | 11 | 26 | 14

BASELINE CHARACTERISTICS:
Population: Four subjects from safety set who had no post-baseline OFF-time efficacy assessment were excluded from the full analysis set: three (1.9%) subjects in the OPC 50 mg group and one (0.7%) subject in the placebo group.
Groups:
- Total: Total of all reporting groups
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | Placebo | Total
Number analyzed (Participants) | 125 | 147 | 135 | 407
Age, Customized [Number; unit: participants]
  <70 years | 96 | 96 | 107 | 299
  ≥70 years | 29 | 51 | 28 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 89 | 71 | 242
  Male | 43 | 58 | 64 | 165

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of 2 BIA 9-1067 (25 mg, and 50 mg) Compared With Placebo, When Administered With the Existing Treatment of L-DOPA Plus a DDCI (DOPA Decarboxylase Inhibitor)
Description: Efficacy of 2 BIA 9-1067 (25 mg, and 50 mg) compared with placebo, when administered with the existing treatment of L-DOPA plus a DDCI (DOPA decarboxylase inhibitor), in patients with PD and end-of-dose motor fluctuations. The primary efficacy variable will be the change from baseline in absolute OFF-time at the end of the DB period.
Time Frame: 14-15 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | Placebo
Number analyzed (Participants) | 125 | 147 | 135
minutes | -102.8 (159.42) | -124.0 (178.23) | -64.5 (155.35)

2. Secondary Outcome: UPDRS (Unified Parkinson's Disease Rating Scale) Sections I (ON), II (ON and OFF), and III (ON)
Description: Total UPDRS SCORE (I, II (ON), and III) Change from Baseline to Endpoint
  * UPDRS I evaluation of mentation, behavior, and mood
  * UPDRS II self-evaluation of the activities of daily life (ADLs) including speech, swallowing, handwriting, dressing, hygiene, falling, salivating, turning in bed, walking, and cutting food
  * UPDRS III clinician-scored monitored motor evaluation The UPDRS I, II and III scores and subscores are calculated as the sum of all individual items. If one or two items in a scale are missing, they will be imputed with the mean of the non-missing items of that scale.
  Subscale has 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe
  The final cumulative score will range from 0 (no disability) to 199 (total disability).
Time Frame: 14-15 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | Placebo
Number analyzed (Participants) | 125 | 147 | 135
units on a scale
  Baseline | 30.8 (16.88) | 31.7 (17.55) | 31.5 (17.00)
  Endpoint | 26.6 (16.40) | 28.7 (18.11) | 28.1 (16.78)

3. Secondary Outcome: Parkinson's Disease Sleep Scale (PDSS)
Description: The Parkinson's disease Sleep Scale (PDSS) is a specific scale for the assessment of sleep disturbances in subjects with PD. The PDSS score is calculated as the sum of all single items. If one or two items are missing, they will be imputed with the mean of the non-missing items. If three or more items are missing, no imputation will be done and the score will be set to missing.
  Subscale has 0-10 ratings, where 0 = severe and 10 = normal
  The PDSS total score is a sum score of all 15 questions and ranges from 0 to 150, with lower scores meaning more disability.
Time Frame: 14-15 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | Placebo
Number analyzed (Participants) | 123 | 147 | 135
units on a scale
  Baseline | 95.75 (28.026) | 102.62 (25.116) | 101.76 (26.729)
  Visit 5 | 97.99 (26.196) | 103.05 (26.437) | 107.11 (26.987)
  Visit 7 | 98.79 (25.280) | 103.25 (26.752) | 105.39 (28.643)

4. Secondary Outcome: Non-motor Symptoms Scale (NMSS)
Description: The Non-motor Symptoms Scale (NMSS) consists of 30 questions, covering 9 dimensions, whereby each item is scored for severity and frequency: Severity None 0 Mild (symptoms present but causes little distress) 1 Moderate (some distress or disturbance to subject) 2 Severe (major source of distress or disturbance to subject) 3
  Frequency Rarely (<1/wk) 1 Often (1/wk) 2 Frequent (several times per week) 3 Very Frequent (daily or all the time) 4
  The product of frequency and severity is calculated for each item and each dimension score is defined as the sum of the frequency*severity of the respective items. If frequency or severity of a single item is missing, the domain score will not be calculated. The NMSS total score is defined as the sum of all domain scores.
  The NMSS total score is calculated by adding all domain scores (0-360), and lower scores mean less disability.
Time Frame: 14-15 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | Placebo
Number analyzed (Participants) | 125 | 147 | 135
units on a scale
  Baseline | 38.2 (29.40) | 36.7 (30.88) | 38.2 (33.37)
  Visit 5 | 33.7 (26.30) | 33.2 (27.95) | 33.5 (31.18)
  Visit 7 | 35.0 (29.88) | 31.5 (28.47) | 31.6 (29.88)

ADVERSE EVENTS:
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/125 | 9/150 | 5/136
Other Adverse Events (participants affected / at risk) | 87/125 | 108/150 | 68/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 25 mg (N=125) | BIA 9-1067 50 mg (N=150) | Placebo (N=136)
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 0 | 1
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
BIOPSY PROSTATE (Investigations) | 0 | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
COGNITIVE DISORDER (Nervous system disorders) | 0 | 0 | 1
DYSKINESIA (Nervous system disorders) | 1 | 0 | 0
DELIRIUM FEBRILE (Psychiatric disorders) | 0 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 0 | 0
CYSTOCELE (Reproductive system and breast disorders) | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 25 mg (N=125) | BIA 9-1067 50 mg (N=150) | Placebo (N=136)
Dyskinesia (Nervous system disorders) | 30 | 36 | 11
Constipation (Gastrointestinal disorders) | 12 | 10 | 2
Dry mouth (Gastrointestinal disorders) | 13 | 6 | 1
Blood CPK increased (Investigations) | 5 | 12 | 5
Parkinson's disease (Nervous system disorders) | 9 | 6 | 7
Fall (Injury, poisoning and procedural complications) | 7 | 7 | 9
Hypertension (Vascular disorders) | 8 | 6 | 3
Nausea (Gastrointestinal disorders) | 8 | 5 | 8
Headache (Nervous system disorders) | 6 | 6 | 9
Insomnia (Psychiatric disorders) | 10 | 2 | 3
Urinary tract infection (Infections and infestations) | 3 | 9 | 2
Dizziness (Nervous system disorders) | 4 | 6 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1
Somnolence (Nervous system disorders) | 6 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other